CLINICAL TRIAL: NCT06206148
Title: Comparison of Methods for Recording Post Operative Pain: A Prospective Randomized Trial
Brief Title: Comparison of Methods for Recording Post Operative Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 23-40666
Record Dates: First submitted 2024-01-04; First posted 2024-01-16 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Pain, Postoperative
Keywords: Pain Recorder; Device; Self-report
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Post-operative orthopedic surgery patients will be randomly assigned to one of three pain collection methods and instructed to record their pain level as often as they like. The three methods of pain collection are: a hand-written pain journal, a smartphone app, and a novel electronic pain recorder device.
Masking Description: The three different methods are very apparent and masking wouldn't provide any benefit
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Hand-written pain journal (Experimental): Post-operative orthopedic surgery patient will be given a pen and journal with chart inside and instructed to fill out the chart with time/date and pain intensity level as frequently as they want.
  Interventions: Other: Given Hand-written pain journal
- Smartphone app (Experimental): Post-operative orthopedic surgery patient will be given a research smartphone and an app to record their pain and will be instructed to fill out the pain survey as frequently as they want.
  Interventions: Other: Smartphone app
- Novel electronic pain recording device (Experimental): Post-operative orthopedic surgery patient will be given a pain recording device and will be instructed to input their pain using the buttons on the device as frequently as they want.
  Interventions: Device: Given novel electronic pain recording device

INTERVENTIONS:
Device: Given novel electronic pain recording device — Patients in this arm will be given a custom-built pain recording device to see if the method of self-reported data collection has any effect on how many data points are collected.
  Arms: Novel electronic pain recording device
Other: Given Hand-written pain journal — Patients in this arm will be given a hand-written pain journal to see if the method of self-reported data collection has any effect on how many data points are collected.
  Arms: Hand-written pain journal
Other: Smartphone app — Patients in this arm will be given a research smartphone with survey app to see if the method of self-reported data collection has any effect on how many data points are collected.
  Arms: Smartphone app

SUMMARY:
The purpose of the current study is to identify the optimal method of collection of pain intensity data. The study will compare three collection methods: a hand-written pain journal, a smartphone app, and a novel electronic pain recorder device. Patients will be randomly assigned to one of three methods and instructed to record their pain level as often as they like. The number of pain intensity recordings per day will then be compared across groups.

DETAILED DESCRIPTION:
Pain is a universal experience and at the forefront of all things medicine; however, the way medical professionals deal with it lacks coherence. Clinicians often ask their patients how their pain is, but seldom document it with enough information to be useful. The purpose of this study is to determine how we can collect the most self-reported pain intensity data. The investigators will collect this data with time and date-stamped Visual Analogue Scale-a pain rating scale from 0-10-scores for each patient in the study, randomized to one of three groups (pen & paper, app, and pain recorder device). As pain is a universal experience and a hallmark sign of many disease states, having a detailed recording of the patient's pain journey is of utmost importance, and understanding that pain with further granularity can only help with the diagnosis of worsening disease, personalization of treatment, and outcomes assessment.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years old

Exclusion Criteria:

* Patient cannot use a smartphone
* Patient cannot use his hands to write or press a button
* Patient has a nerve catheter (has no pain)
* Altered mental status
* Neuropathy causing loss of pain sensation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 147 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Comparing Methods for Pain Score collection | On patient discharge, up to 2 weeks
  Pain Scores will be measured on the Visual Analog Scale (VAS) via 3 different methods to determine the best way to collect pain intensity data. The Visual Analog Scale goes from 0-10 where 0 means no pain and 10 means maximum pain.

CONTACTS AND LOCATIONS:
Overall Officials: Meir T Marmor, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- Zuckerberg San Francisco General Hospital, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No
Not sharing IPD